CLINICAL TRIAL: NCT04431765
Title: Evaluation of Desensitization Therapy and Re-treatment of Eye Movement Information [EMDR] in Patients With Post-traumatic Stress Disorder [PTSD]: Neuronal Correlates and Cognitive Impact on the Attention and Memory of Emotional Stimuli.
Brief Title: Evaluation of Desensitization Therapy and Re-treatment of Eye Movement Information [EMDR] in Patients With Post-traumatic Stress Disorder [PTSD]
Acronym: ICE-EMDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Januel, Head of the clinical research department (psychiatrist), Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10477M-ICE-EMDR
Record Dates: First submitted 2020-04-30; First posted 2020-06-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Eye Movement Information- Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: In one hand, Patients with Post-traumatic Stress Disorder who will receive Eye Movement desensitization reprocessing therapy and in other hand patient with post-traumatic Stress Disorder who will receive Trauma-Centred Cognitive and Behavioural Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient for Eye Movement desensitization Reprocessing therapy (Active Comparator): Patient with post-traumatic Stress Disorder will receive Eye Movement Desensitization reprocessing therapy
  Interventions: Other: Eye Movement Desensitization Reprocessing therapy
- patients for Trauma-Centred Cognitive and Behavioural Therapy (Placebo Comparator): Patients with post-traumatic Stress Disorder will receive Trauma-Centred Cognitive and Behavioural Therapy
  Interventions: Behavioral: Trauma-Centred Cognitive and Behavioural Therapy

INTERVENTIONS:
Other: Eye Movement Desensitization Reprocessing therapy — The Eye Movement Desensitization Reprocessing therapy uses bi-alternating (right-left) sensory stimulation through eye movements. The patient follows the therapist's fingers from right to left in front of his eyes and also by auditory stimuli. The patient wears a helmet that alternately makes him hear a sound to the right, then to the left or touch the patient holds in his hands buzzers that alternately vibrate from right to left, or alternatively the therapist taps the patient's knees or the back of his hands.
  Other Names: EMDR
  Arms: Patient for Eye Movement desensitization Reprocessing therapy
Behavioral: Trauma-Centred Cognitive and Behavioural Therapy — A CBT is a short, scientifically validated therapy that focuses on the interactions between thoughts, emotions and behaviours. These therapies focus on the current problems of the person, while taking into account their historical causes. They help gradually overcome disabling symptoms and aim to strengthen adaptive behaviours. A CBT relies on different techniques that help the patient to identify the mechanisms at the origin of his difficulties, to experiment with new behaviors and thus to gradually come out of vicious circles that perpetuate and aggravate the psychic suffering.
  Other Names: CBT
  Arms: patients for Trauma-Centred Cognitive and Behavioural Therapy

SUMMARY:
This research aims to confirm that the therapeutic effect of EMDR is associated with changes in the interaction between cognitive function and emotional stimuli in PTSD patients compared to a controlled therapy in a randomized, single-blind study.On the other hand, this study aims to observe neuronal and cognitive correlates related to EMDR therapy compared to a control therapy.

This investigation would improve the understanding of the mechanisms of action of the EMDR, still unknown to date.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with PTSD according to DSM 5 criteria (APA 2013) related to a single traumatic event,
* Aged 18 to 65 years,
* Signed informed consent.
* Patient with social security affiliation or State Medical Aid (AME)

Exclusion Criteria:

* Neurological disorders
* No other major psychiatric disorders than PTSD (DSM 5)
* Severe and/or unstable somatic pathologies,
* Patient not affiliated with social security,
* Patient hospitalized under stress in psychiatric care at the decision of the state representative or in psychiatric care at the request of a third party,
* Patient under guardianship,
* Patient participating in parallel with other biomedical research,
* Change of antidepressant during the last three months,
* Patient not fluent in French
* MR-specific criteria for not inclusion:
* women of childbearing age without effective contraception or a positive pregnancy test,
* patients carrying pacemakers or electrical or electronic devices, clips or metal prostheses,
* subjects with neurological disorders, cerebral abnormalities or suffering from claustrophobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Post Traumatic Stress Scale-5 (PCL-5) | Before the therapy begins, at day 0
  The PCL-5 is a self-assessment consisting of 20 items that measures the 20 PTSD symptoms of the DSM-5. The wording of the PCL-5 items reflects both changes in existing symptoms and the addition of new symptoms in the DSM-5.
  The objectives of PCL-5 are numerous, such as monitoring changes in symptoms during and after treatment, screening individuals with PTSD, making an interim diagnosis of PTSD.
Post Traumatic Stress Scale-5 | Within 3 weeks before the end of the therapy
  The PCL-5 is a self-assessment consisting of 20 items that measures the 20 PTSD symptoms of the DSM-5. The wording of the PCL-5 items reflects both changes in existing symptoms and the addition of new symptoms in the DSM-5.
  The objectives of PCL-5 are numerous, such as monitoring changes in symptoms during and after treatment, screening individuals with PTSD, making an interim diagnosis of PTSD.
State Trait Anxiety Inventory (STAI) | Before the therapy begins, at day 0
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.
State Trait Anxiety Inventory (STAI) | Within 3 weeks before the end of the therapy
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety.
The Short Form (36) Health Survey (SF36) | Before the therapy begins, at day 0
  TheSF36isashortquestionnairewith36itemswhichmeasureeightmulti-itemvariables:physicalfunctioning(10items),socialfunctioning(twoitems),rolelimitationsduetophysicalproblems(fouritems),rolelimitationsduetoemotionalproblems(threeitems),mentalhealth(fiveitems),energyandvitality(fouritems),pain(twoitems),andgeneralperceptionofhealth(fiveitems).Foreachvariableitemscoresarecoded,summed,andtransformedontoascalefrom0(worstpossiblehealthstatemeasuredbythequestionnaire)to100(bestpossiblehealthstate).
The Short Form (36) Health Survey (SF36) | Within 3 weeks before the end of the therapy
  TheSF36isashortquestionnairewith36itemswhichmeasureeightmulti-itemvariables:physicalfunctioning(10items),socialfunctioning(twoitems),rolelimitationsduetophysicalproblems(fouritems),rolelimitationsduetoemotionalproblems(threeitems),mentalhealth(fiveitems),energyandvitality(fouritems),pain(twoitems),andgeneralperceptionofhealth(fiveitems).Foreachvariableitemscoresarecoded,summed,andtransformedontoascalefrom0(worstpossiblehealthstatemeasuredbythequestionnaire)to100(bestpossiblehealthstate).
Childhood Trauma Questionnaire (CTQ) | Before the therapy begins, at day 0
  The Childhood Trauma Questionnaire (CTQ) is a questionnaire developed by Bernstein et al. (1994) that includes 70 items with a Likert scale in five response choices (from 1 = "never true" to 5 = "very often true").
Childhood Trauma Questionnaire (CTQ) | Within 3 weeks before the end of the therapy
  The Childhood Trauma Questionnaire (CTQ) is a questionnaire developed by Bernstein et al. (1994) that includes 70 items with a Likert scale in five response choices (from 1 = "never true" to 5 = "very often true").
Clinician Administered PTSD Scale for DSM-5[CAPS-5]) | Before the therapy begins, at day 0
  he CAPS-5 is a 30-item structured interview that can be used to:
  Make current (past month) diagnosis of PTSD,Make lifetime diagnosis of PTSD, Assess PTSD symptoms over the past week
Clinician Administered PTSD Scale for DSM-5[CAPS-5]) | Within 3 weeks before the end of the therapy
  he CAPS-5 is a 30-item structured interview that can be used to:
  Make current (past month) diagnosis of PTSD,Make lifetime diagnosis of PTSD, Assess PTSD symptoms over the past week
Clinical Global Impression (CGI) | Before the therapy begins, at day 0
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders
Clinical Global Impression (CGI) | Within 3 weeks before the end of the therapy
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Januel, MBBS, Principal Investigator — CHVille Evrard
Locations (1):
- Ch Ville Evrard, Neuilly-sur-Marne, France